CLINICAL TRIAL: NCT05995873
Title: A Project to Test the Efficacy and Safety of An Innovative Treatment for Opiate Use Disorders.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MindLight, LLC (Industry)
Collaborators: Mclean Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R44DA050358 (NIH)
Record Dates: First submitted 2023-07-14; First posted 2023-08-16 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-08

CONDITIONS: Opioid Use Disorder, Moderate; Opioid Use; Opioid Dependence; Opioid Abuse; Opiate Dependence; Opioid Use, Unspecified
MeSH Terms: conditions — Opioid-Related Disorders; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: 130 participants will be treated with unilateral transcranial photobiomodulation to their brain hemisphere with a more positive emotional valence. Half will receive sham and half active. Treatment will be 2 times a week for 4 weeks, then once a week for 20 weeks and then a followup 1 week later. The study will be half at MindLight, LLC and half at McLean Hospital.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only the treater knows whether the participant receives the sham or active treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- treatment (Sham Comparator): Half of the participants will receive sham. Treatment will be 2 times a week for 4 weeks, then once a week for 20 weeks and then a followup 1 week later. The sham device is identical to the active device except that it has foil over the LED.
  Interventions: Device: unilateral transcranial photobiomodulation
- Active treatment (Experimental): Participants in this group will receive a 4-minute unilateral transcranial photobiomodulation treatment.
  Interventions: Device: unilateral transcranial photobiomodulation

INTERVENTIONS:
Device: unilateral transcranial photobiomodulation — An 810nM LED at 240mW/cm2 is placed at either F3 or F4 for 4 minutes.

SUMMARY:
Investigators will test, for safety and efficacy, a novel treatment for opiate addiction that applies a 4-minute treatment of intense near infra-red light to stimulate a side of the brain that the investigators determine to be healthier, more mature, and less traumatized. Investigators will compare among actively using participants an active and a sham treatment given either once or twice weekly for 25-weeks at 2 sites. Investigators hope this will lead to a significant weapon in the battle against the opioid epidemic as well as lead to psychological and physiological insights into possible relations among trauma, cerebral laterality, and addiction.

DETAILED DESCRIPTION:
Approach. Investigators have had a and productive Pre-submission meeting with the FDA on April 21, 2022, and are following their guidance in our approach. The goal of this Phase II study is to test further the efficacy and safety of a new and innovative, patented application of transcranial photobiomodulation for the treatment of opioid use disorder (defined by DSM-5 criteria) with the possibility of achieving FDA clearance. The Opioid Addiction Therapy System is a photobiomodulation device platform intended to be used alone or as an aid to psychotherapy and medical-assisted treatments to treat opioid use disorder. It is intended to be used by trained psychotherapists in clinical environments on patients with opioid use disorder.

Specific Aim1:

1. Following FDA's preliminary guidance, Investigators aim first to assess whether active Rx with UtPBM administered to the more positive hemisphere helps participants taper and abstain from use of opioids as indicated by an increase in the percent of weekly visits in which there was no self-reported use of opioids on TimeLine Follow Back and urine screens for opioids were negative. This will be assessed from weeks 10 through 26, to give participants sufficient time to taper off opioids. An additional primary outcome will be the reduction in frequency of use (days per week) as assessed using timeline feedback from baseline to week 26. Secondary outcome measures will include the following: retention in treatment, opioid craving, withdrawal symptoms, clinical global impression ratings of severity and improvement, quality of life metrics and Treatment Success, as at least 80% opioid abstinence during weeks 10-26. An assessment will also be made of adverse events during the treatment period.

   Milestones: a. Investigators predict based on our Phase I findings that active treatment will increase weekly abstinence rates by 20% or more over sham treatment (e.g., 30% vs 10% weekly opioid-negative visits). Investigators expect each of the secondary outcomes to be significantly better in the active group with a p value of less than 0.05.
2. Investigators wish to see if actively treated participants age more slowly over the 26-week course of the study than those who receive the sham treatments. Investigators will measure this by using epigenetic techniques. Investigators will use state-of-the-art epigenetic measures of Intrinsic Epigenetic Age Acceleration to assess subtype differences in DNA m. Investigators feel this is superior focusing on candidate genes. Peripheral lymphocytes are the most appropriate cell type for assessing Intrinsic Epigenetic Age Acceleration.

Sequence of Visits. Interested individuals will call to receive information and will complete a brief screen for age and key exclusion criteria. Those who appear eligible will be invited to interview. Visit 1 will consist of full study informed consent, structured interviews to assess inclusion and exclusion criteria, TimeLine Followback to assess current degree of substance use, urine drug screen and computerized assessment of hemispheric emotional valence. Those who meet entrance criteria and agree to participate will be randomized into active or sham groups. Treatment sessions will start with visit 1 and will occur twice weekly for 6 weeks, then weekly until week 25 with one untreated follow-up session on week 26.

Within Session Protocol. Participants will give verbal reconsent to be in the study at each study session. Immediately before each UtPBM active and sham treatment, the primary and the secondary outcome measures will be recorded.

The active treatment will consist of applying PBM in the form of a super-luminous LED with an output of 250 mW/cm2 at a frequency of 810 nM with a width of 40 nM when applied the skin for a fluence of 60J/cm2. The treatment will consist of the exposure to the light for 4 minutes at one of 2 sites on the forehead that correspond to the 10-20 electroencephalogram sites, F3, and F4. Whether Investigators will treat at F3 or F4 will be determined by the tests of HEV. Investigators will treat the side that is determined to have a more positive HEV. Based on a penetration of 3.7% of the light to the dura, Investigators will be applying 2.1 Joules/ cm2 to the treated area of the brain. Our level of light exposure is well below the ANSI standard of 0.32 W/cm2. The fluence of our device is 40 times less than the device that was used in the study of 1410 stroke patients without any observed side-effects and was found in a study of the rat brain exposed to light to cause no observable behavioral or cellular alterations. The device has been determined by the FDA to be of no significant risk as described in the attached FDA letter of September 8, 2022.

The sham treatment will be identical to the active treatment except that the LED will be covered with aluminum foil to prevent near-infrared light from reaching the brain. The treating clinician, who will not be blinded, will apply the either the active or the sham treatment to the participant in a manner that does not allow either the recording clinician or the patient to have any way to detect whether a given treatment is active or sham. When asked in prior studies, neither the patients nor recorders were able to detect whether the application was active or sham at the time of treatment.

Although Investigators believe that the procedures in this study are not expected to cause adverse effects, during all procedures the researcher in attendance will closely observe the subject for any adverse effects. All NIH and WCG IRB patient safety and monitoring procedures will be followed. For any adverse events Investigators will use the NIH Adverse Events Form. All serious adverse events will be report to the IRB, NIH and FDA and posted to clinicaltrials.gov.

Subjects will not wear protective eyewear. The researcher administering the tPBM will be careful to not shine the LED into the subjects' eyes. LEDs do not pose the level of danger to the eyes that lasers present because the LED light is not coherent; still a person's staring into a super-luminous LED for 4-minutes could potentially cause damage the eye, but a second or two of looking at the LED will not cause harm. Photobiomodulation is currently used to treat some retinal diseases.

Any subject who for any reason wishes to leave the study at any time before its conclusion, of course, will be free to do so. If any unexpected, unacceptable adverse events are observed, Investigators will discontinue the entire study until Investigators have fully consulted with the IRB.

Each session will include use assessment of frequency and extent of opioid and other substances, urine analysis with temperature check for drug use, pregnancy testing of female participants, assessment of hemispheric emotional valence, symptom ratings and active or sham UtPBM. Following treatment, participants who revealed drug use, or had a positive urine assay, will be provided with instructions on how to safely taper opioid use (e.g., 10-20% reduction per week if using daily, discontinuation if using less frequently). Participants who have reduced intake from baseline will also be cautioned at each visit that there is an increased risk for overdose if they abruptly return to a previously used higher dose as it can take as little as a week to lose tolerance.

Investigators have extensive experience with our device and method and in clinical practice and in a study, Investigators intentionally activated the negative hemisphere, and this can cause the patient to feel his usual anxiety and symptoms but has never created a danger. All treating personnel are well trained in our techniques. Investigators will not blame a failure to reach our milestones on treatment of the wrong side; Investigators are testing our method of determining the side of the greater HEV and treating it.

Outcome Measures: Primary Measure of efficacy will be percent abstinence from opioid use, defined as the percent of each participant's weekly visits that are negative for opioid use both on the use report and by urine analysis from weeks 10-26. If a participant misses a visit, Investigators will attempt to contact them by phone for a use rating and to have them provide a urine sample at a test center. Otherwise, all missed samples or ratings will be defined as non-negative. In addition, Investigators will also assess whether there was a significant difference between active and sham treatment in the frequency (days per week) of use based on the use report, which Investigators have found in our studies to reveal a greater degree of use than once or twice weekly urine tests, and which provides more granularity than designating each week (or test) as positive or negative. This is the approach that Investigators used to analyze opioid use from the phase I study and makes sense as the proposed protocol does not include a detoxification stage.

Secondary Measures include the following standard outcome measures: retention in treatment, opioid craving, withdrawal symptoms, clinical global impression ratings of severity and improvement, and Treatment Success, as at least 80% opioid abstinence during weeks 10-26. Secondary outcomes have been used in one or more of the RCTs designed to test the efficacy of buprenorphine for opioid use disorder. Investigators will also include visual analog scale ratings of quality of life and quality of relationships and the Hamilton Depression Rating Scale and the Hamilton Anxiety Rating Scale.

Opioid craving will be assessed using the Opioid Craving Visual Analog Scale (0-100 mm). Withdrawal symptoms will be assessed using the Clinical Opioid Withdrawal Scale. Investigators will also use the Subjective Opiate Withdraw Scale and the Columbia Suicide Severity Scale. Retention will be assessed as the number of sessions attended as determined by their discontinuation or removal. Participants will be removed from the study if they engage in a dangerous or sexually inappropriate manner with staff or have a positive pregnancy test. Investigators will conduct analyses of both discontinuation, which will include all participants who fail to complete the full trial, and a specific analysis of the voluntary drop-out rate that would include participants who exit the study, are lost to follow up, receive medication assisted treatment or other somatic modalities, but would exclude legitimate unavoidable reasons for discontinuation such as pregnancy, parole violation or verifiable illness or injury unrelated to current opioid use disorder that would preclude participation.

Investigators will measure Intrinsic epigenetic age acceleration using the whole methylome chip. For these analyses, Investigators will use the EWAS of that provides an epigenetic measure of low-grade chronic inflammation from an additive weighted score of 58 replicated CpG sites in European and African-Ancestry samples. Intrinsic epigenetic age acceleration will be assessed from the Epic Methylome array. This parameter typically correlates highly with chronological age, however, emerging evidence from our lab and others point to an acceleration of epigenetic aging in response to cumulative lifetime stress, childhood maltreatment, and post-traumatic stress disorder. All saliva samples will be stored and processed at McLean Hospital which has specimen and data security in place.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant females between 18-65 years of age
* Individuals having an opioid use disorder with mild-to-moderately severe symptoms

Exclusion Criteria:

* Individuals who are pregnant,
* Individuals who are psychotic,
* Individuals who are actively suicidal,
* Individuals who are a danger to self or others,
* Individuals who are who have a history of severe psychiatric or neurological disorders or life-threatening medical illness.
* Individuals will be excluded with chronic pain requiring opioid treatment.
* Individuals who are who are breastfeeding,
* Individuals who are adults requiring a legally authorized representative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
percent of participants that achieve abstenense | up to 26 weeks
  we will test for use with urine and hair test

SECONDARY OUTCOMES:
Overall clinical status | at the end of the study
  Clinical Global Impressions Scale

CONTACTS AND LOCATIONS:
Locations (1):
- MindLight, LLC, Newton Highlands, Massachusetts, United States

REFERENCES:
- [Background] Schiffer F, Khan A, Bolger E, Flynn E, Seltzer WP, Teicher MH. An Effective and Safe Novel Treatment of Opioid Use Disorder: Unilateral Transcranial Photobiomodulation. Front Psychiatry. 2021 Aug 10;12:713686. doi: 10.3389/fpsyt.2021.713686. eCollection 2021. PMID 34447323
- See also: Article: An Effective and Safe Novel Treatment of Opioid Use Disorder — https://www.frontiersin.org/articles/10.3389/fpsyt.2021.713686/full